CLINICAL TRIAL: NCT02427100
Title: Evaluation of a Shelter-Based Diet and Physical Activity Intervention for Homeless Adults: A Pilot Study
Brief Title: Evaluation of a Shelter-Based Diet and Physical Activity Intervention for Homeless Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other); American Cancer Society, Inc. (Other); Simmons Cancer Center (Other)
Responsible Party: Principal Investigator, Darla Elizabeth Kendzor, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU 062014-031
Record Dates: First submitted 2014-12-17; First posted 2015-04-27 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-02

CONDITIONS: Dietary Modification; Physical Activity
Keywords: Homeless; Randomized Controlled Trial; Diet; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Control participants will be paid for assessments. They will receive study newsletters and a pedometer with advice after the final follow-up visit.
- Intervention Group (Active Comparator): Intervention participants will receive 4 weekly newsletters, a pedometer with walking advice, and twice daily fruit/vegetable snacks during weekdays.
  Interventions: Behavioral: Diet/Physical Activity

INTERVENTIONS:
Behavioral: Diet/Physical Activity — Diet/Physical Activity Intervention
  Arms: Intervention Group

SUMMARY:
The proposed study will utilize a randomized controlled trial design to pilot-test a 4-week shelter-based diet and physical activity intervention in a sample of homeless adults residing in the transitional shelter at The Bridge Homeless Assistance Center in Dallas, TX (N = 50). Participants will be randomly assigned to a diet/physical activity intervention group (n = 25) or a paid assessment-only control group (n = 25). Three intervention strategies will be employed: 1) computer-tailored newsletters adapted from a program supported for use in other populations, 2) the distribution of fruit and vegetable snacks directly to individuals, and 3) the provision of pedometers and walking goals. Thus, the primary aim of the proposed study is to 1) evaluate the feasibility and effectiveness (relative to an assessment-only control group) of a shelter-based intervention designed to improve dietary intake and increase physical activity among homeless individuals. The main study outcomes will be average daily fruit and vegetable consumption and objective pedometer/ accelerometer assessment of physical activity (assessed weekly) over the 4-week study period, and at a follow-up assessment 4 weeks after the conclusion of the intervention. Secondary aims will focus on: 2) identifying intervention-related differences (relative to the control group) in indicators of physical health including blood pressure, weight, body mass index (BMI), waist circumference, and other dietary variables (i.e., caloric intake, meals consumed outside of the shelter, daily fat and fiber intake) and 3) identifying psychosocial variables associated with dietary quality and physical activity.

DETAILED DESCRIPTION:
Study Overview. The proposed study will take place at "The Bridge" homeless shelter in Dallas, TX. The study intervention will use a randomized controlled trial design, and an additional 50 transitional shelter residents will be recruited to participate in the proposed 8-week study (4-week intervention; 4-week post-intervention follow-up visit). Transitional Shelter residents stay in "semi-private" rooms for an average of 5 months while staff works to secure more permanent housing. Interested and eligible participants will be randomized to either 1) a 4-week shelter-based diet or physical activity intervention, or 2) standard care (paid assessment only). Participants will be asked to complete weekly assessments of diet, physical activity, stress, readiness to change, and other relevant variables throughout the 4-week intervention period, in addition to a 4-week post-intervention follow-up. Participants will be compensated with gift cards for each of 6 visits. Participants assigned to the control group will receive tailored newsletters and pedometers with walking goals at the final follow-up visit. Laptop and tablet computers equipped with Questionnaire Development System software will be transported to the shelter for all intervention and assessment sessions.

Intervention Components Education. A series of four computer-tailored newsletters will be generated for each individual participant using TailorTool, a web-based program hosted and maintained at the University of North Carolina (described below; see also www.chaicore). Newsletter topics include healthy eating (especially the importance of fruit/vegetable consumption), physical activity, and weight management. Using information collected at baseline, newsletters will be tailored to individual participants based on demographic, psychosocial, behavioral, and community resource information. The program will be adapted to include graphics and testimonials relevant to the sheltered homeless population. Strategies for healthy food selection and community resources available to shelter residents will be provided.

The newsletters will include of a set of tailored "stories" in the following formats designed to appeal to the homeless shelter population: Testimonials (tailored to gender) by residents of the shelter who have made changes in weight and lifestyle. An advice column (tailored to behavior-specific barriers), that uses a "Dear Abby" format in which an expert (e.g., dietician) answers questions tailored to participant-selected barriers. Behavioral feedback (current behavior compared to recommendations) will be provided. Stage of change-based action plan (tailored to stage of change, current behavior) will offer a specific set of steps that are stage-matched to participant readiness to change related to each behavior. The importance of social support (tailored to behavior-specific social support/network characteristics) will be discussed by providing a targeted story about how social support (tailored to type of support and person most helpful to give support) has helped someone make healthy changes. The values section (tailored to participant-selected core values) discusses the participant-selected values and suggests possible ways that these values may be related to the target behavior. Community resources will provide information and tips tailored to the shelter, such as group session information, healthful choices in the cafeteria (and other common food sources), maximizing SNAP food benefits for optimal nutrition, good nutrition with a limited income, walking groups, contact information, and community resources. Participants assigned to standard care will receive the tailored newsletters after they complete the final follow-up assessment.

TailorTool is a software tool created by the UNC CHAI (Communication for Health Applications and Interventions) Core that enables the creation and delivery of tailored communications in a dynamically generated pdf newsletter format. The tool generates intervention material such as individual feedback on targeted behavior(s) and variables such as relevant demographics, psychosocial factors, and barriers. Templates of various page lay-out possibilities allow individualization of the look of the newsletters. Messages are drawn from a message library of text files of varying lengths depending on the needs of the research study. Graphics can be imported into the various template pages. Newsletters can vary in length and can be personalized with names of participants. Following completion of an online survey the newsletter(s) are created in a pdf format for reading, saving, and/or printing by the participant. Each subsequent newsletter can be available immediately or timed for release to fit the timeline of the intervention.

From a technical perspective, the web application for the automated web-to-print system is programmed to run under a Windows operating system, using open-source software and a MS SQL database. The core of the system is a server-side application, with the website consisting of ASP pages (Active Server Pages), which interface with the application using XML. The backend application is heavily database-driven with everything from survey questions and skip patterns (i.e. which survey answers can cause later questions to be disabled, as described above; the actual disabling takes place client-side, with dynamically-generated javascript code) to the newsletter content and tailoring logic stored in, and thus configurable via, XML files. Participants' survey-response data are stored in the database. The dynamic generation of the print newsletters in pdf format is done within the application using a dynamic-link library installed on the system.

Fruit/Vegetable Snacks. We will provide transitional shelter residents assigned to the intervention group with two pieces of fruit and/or vegetables each weekday. We will offers fruits/vegetables that are easy to distribute and do not require preparation other than washing or packaging in a bag (e.g., apples, bananas, oranges, baby carrots, broccoli, cauliflower). Foods will be purchased by study staff, stored at The Bridge in the cafeteria refrigerator, and offered to participants assigned to the intervention group in the cafeteria at specified times twice daily as mid-morning and mid-afternoon snacks. Note that because the snacks will be offered between regular mealtimes, only intervention participants will be in the cafeteria to receive the fruit/vegetable snacks. In addition, snacks will be consumed in the cafeteria during specified snack times because the shelter does not allow food in other areas of the building. Study staff will follow all relevant shelter food safety practices. It is hypothesized that study participants will consume more fruit and vegetables and eat fewer meals/snacks from fast food restaurants and convenience stores than individuals assigned to the control group. This is a practical, simple, and direct approach to increasing fruit/vegetable consumption, as shelter residents obtain most of their meals from the shelter and offering snacks may discourage residents from seeking less healthful foods elsewhere.

Pedometers. Walking is a practical way to achieve physical activity recommendations among individuals experiencing homelessness, as it does not require any specific equipment and may be a common activity and means of transportation in this population. Pedometers are small and inexpensive devices that measure steps walked per day. All study participants will be provided with a New Lifestyles NL-1000 pedometer/ accelerometer, which measures steps, distance, and activity minutes and is equipped with a 7-day memory and clock. Those randomly assigned to the intervention will be instructed to aim for 10,000 steps per day, but to focus on gradually increasing their steps each day (rather than achieving 10,000 steps right away) if they are currently very sedentary. In addition, intervention participants will be provided with information about the Back on My Feet program, which is offered at the Bridge shelter. Program members meet for a group run/walk 3 times per week on Monday, Wednesday, and Friday mornings. Intervention participants will be instructed to wear their pedometer during waking hours each day, and asked to return each week over a 4-week period (4 visits total) so that study staff may record the daily step counts. We will additionally ask participants to return for a 4-week post-intervention follow-up (we will remind participants to wear their pedometer the week prior to the assessment). Individuals assigned to the control group will provided with a pedometer and step goals after the final follow-up visit. All participants may keep their pedometer after their participation in the study is completed. Note that intervention and control group participants will be provided with accelerometers at the beginning of the study to provide an objective measure of physical activity.

ELIGIBILITY:
Inclusion Criteria:

1. at least 18 years of age,
2. willing and able to attend all study visits,
3. earn a score ≥ 4 on the REALM-SF indicating > 6th grade literacy level,
4. physically able to walk and/or run for physical activity,
5. resident of the transitional shelter (must show Bridge ID badge), and
6. have been living in the transitional shelter for ≤ 3 months.

Exclusion Criteria:

1. < 18 years of age,
2. unwilling or unable to attend all study visits,
3. earn a score < 4 on the REALM-SF indicating ≤ 6th grade literacy level,
4. unable to participate in the walking/running component of the intervention (i.e., mobility impairments),
5. are not residents of the transitional shelter (or does not have a Bridge ID badge) or
6. have been living in the shelter for > 2 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darla E. Kendzor, Ph.D., Principal Investigator — The University of Texas Health Science Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to publication — http://journals.humankinetics.com/toc/jpah/0/0

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 15 | 17
Completed | 15 | 15
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.27 (9.88) | 49.35 (6.34) | 48.38 (8.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 9 | 15 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 15 | 27
  White | 1 | 2 | 3
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 17 | 32
BMI, Mean (SD) [Mean (Standard Deviation); unit: kg/m²] | 29.38 (7.27) | 30.20 (7.62) | 29.82 (7.35)
Fruit/Vegetables, cups (past 24 hours) [Mean (Standard Deviation); unit: cups] | 2.60 (1.61) | 3.10 (2.10) | 2.87 (1.87)
Physical Activity Guidelines, n (based on self-report) [Number; unit: participants]
  Not Meeting Guidelines | 8 | 6 | 14
  Meeting Guidelines | 7 | 11 | 18

OUTCOME MEASURES:

1. Primary Outcome: Automated Self-Administered 24-Hour Dietary Recall: Fruit/Vegetable, Cups
Time Frame: 4 weeks post-enrollment
Population: In the control group (n = 15), 1 participant who attended the visit did not complete a dietary recall (leaving a total of 14 participants). In the intervention group, 2 participants did not attend the visit, and 1 who attended did not complete a dietary recall (leaving a total of 14 participants).
Measure: Least Squares Mean (Standard Error); unit: cups
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 14 | 14
cups | 2.08 (.74) | 3.56 (.74)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority or Other; p = .18, ANCOVA

2. Primary Outcome: Accelerometer-Measured Physical Activity: Moderate to Vigorous Intensity Physical Activity
Description: Linear Mixed Model (LMM) methods were used to evaluate differences in daily accelerometer-measured MVPA measured over a 28-day period using SAS version 9.4. Daily accelerometer measured activity was NOT averaged or summarized into a single variable. Rather, daily activity summaries over 28 days were compared between the intervention and control group (see Kendzor et al., 2017, Journal of Physical ACtivity and Health).
Time Frame: Daily over 4 weeks (repeated measures analysis; day 15 excluded because accelerometers were replaced with newly charged accelerometers)
Population: All participants included.
Measure: Median (Inter-Quartile Range); unit: daily minutes
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 15 | 17
daily minutes | 41 [11 to 64] | 60 [28 to 107]
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority or Other; p = .00036, Mixed Models Analysis — The Linear Mixed Model (LMM) regression analysis (repeated measures) was adjusted for daily minutes of accelerometer wear time, gender, age, BMI, education, and meeting physical activity guidelines at baseline; A fourth root transformation of daily accelerometer-measured minutes of MVPA was used to normalize the distribution and was included in the analyses

ADVERSE EVENTS:
Arm/Group | Control Group | Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 0/15 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No